CLINICAL TRIAL: NCT05849675
Title: An fMRI Investigation of the Effects of Selective Histamine-3 Receptor Antagonism on Cognitive and Emotional Processing in Healthy Individuals
Brief Title: Pitolisant Effects on Affect and Cognition Exploratory Study (PEACE Study)
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PEACE
Record Dates: First submitted 2023-04-03; First posted 2023-05-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-03

CONDITIONS: Anhedonia; Cognitive Function
Keywords: Drug; fMRI; pharmaco-fMRI; Cognition; Histamine
MeSH Terms: conditions — Anhedonia | interventions — pitolisant

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups (pitolisant or placebo). This study uses a novel procedure known as variance minimisation (described in Sella, Raz & Cohen Kadosh, 2021) to randomise participants allocation to the two intervention groups based on equalising baseline cognitive functioning and gender. Participants will receive a single dose of the drug (pitolisant, 36mg) or placebo, and undertake fMRI and cognitive/emotional assessment three hours after dose. The study is assessing the effect antagonising the H3 receptor on functional connectivity/cognitive ability, it is not an efficacy or safety study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Matched placebo capsule
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pitolisant (Experimental): Two film-coated tablets (18mg x 2 [36mg]) for oral administration will be encapsulated in an opaque capsule.
  Interventions: Drug: Pitolisant 17.8 MG [Wakix]
- Placebo (Placebo Comparator): Two lactose film-coated tablets (2 x 65mg [125mg]) will be encapsulated in an opaque capsule (identical to the experimental arm drug).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant 17.8 MG [Wakix] — Single dose pitoliosant (36mg)
  Arms: Pitolisant
Drug: Placebo — Single dose placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the effects of selective histamine 3 antagonist pitolisant on brain function and cognition in healthy individuals. The main questions it aims to answer are:

1. Does pitolisant alter functional activity in brain regions linked to reward and cognitive processing during rest or cognitive task performance?
2. Does pitolisant alter cognitive ability across a range of psychological domains, including working memory, executive functioning and emotional processing?

Participants will undertake fMRI scanning in addition to a battery of tasks designed to measure cognitive and emotional processing after taking a single dose of pitolisant or placebo. Researchers will compare differences in functional activity, cognition and emotional processing across the pitolisant and placebo groups.

DETAILED DESCRIPTION:
Cognitive and affective processing are underpinned by monoaminergic neurotransmission and neurosteroid systems, yet there are many aspects of these systems that remain unknown in humans. In particular, monoaminergic histamine 3 (H3) receptors are abundant in CNS regions underpinning cognitive processing (prefrontal cortex, hippocampus, and striatum), yet the role of these receptors in humans remains unclear. Evidence from animal models suggests H3R antagonism improves cognitive functioning, however these specific effects are yet to be examined in humans. Similarly, the function of sigma-1 (σ-1) receptors in the brain is not well understood in humans despite strong evidence of pro-cognitive effects in animal models.

The study will investigate the effect of pitolisant, a dual H3R antagonist and σ-1R agonist, on cognitive and affective processing, in addition to changes in functional connectivity. These effects will be measured with a battery of neuropsychological tasks (e.g., Affective Go/No-Go Task; Adaptive dual n-back task), self-rated measures of cognitive function (PDQ), and resting state fMRI and fMRI data acquisition during the verbal n-back and memory encoding tasks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Not currently taking any medications which may interfere with pitolisant, including psychoactive medications
* Not currently using antihistaminergic medication
* Aged 18-45 years
* Male or female
* Sufficiently fluent English to understand and complete cognitive tasks and questionnaires
* Body Mass Index above or below 18-30
* Right handed

Exclusion Criteria:

* Current pregnancy (as determined by urine pregnancy test taken during screening visit), planning to become pregnant or breast feeding
* Any past or current history of severe and/or serious psychiatric disorder, including but not limited to schizophrenia, psychosis, bipolar affective disorder, major depressive disorder, obsessive compulsive disorder
* Clinically significant abnormal values for urine drug screen, blood pressure measurement ( in accordance with AP20 'non-invasive blood pressure') and ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* History of, or current medical conditions which, in the opinion of the investigator, may interfere with the safety of the participant or the scientific integrity of the study, including epilepsy/seizures, brain injury, hepatic or renal disease, acid-related gastro-intestinal problems, Central Nervous System (CNS) tumours, neurological conditions
* Current or past history of drug or alcohol dependency
* Severe lactose intolerance
* Use of recreational drugs (e.g. cannabis, cocaine, amphetamines) within past 3 months
* Participation in a study which uses the same computer tasks as those in the present study (determined by asking participants about previous studies participated in during screening) within past 3 months
* Participation in a study that involves the use of a medication within the last three months
* Smoking > 5 cigarettes per day
* Consumption of a high amount of caffeine per day (> 400ml caffeine) (e.g., 5 or more cups of coffee)
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator
* Any contraindication to MRI scanning (e.g. metal objects inside the body, pacemakers, significant claustrophobia)
* Not right handed

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
BOLD signal levels during resting state fMRI sequence | 3-6 hours after single dose of drug or placebo.
  Blood Oxygenation Level Dependent (BOLD) signal level in prior regions of interest (striatum, hippocampus and anterior cingulate cortex) in pilosant group compared with the placebo group
BOLD signal levels during fMRI memory encoding task | 3-6 hours after single dose of drug or placebo.
  BOLD signal level in prior regions of interest during the task (hippocampus; perirhinal cortex) in pilosant group compared with the placebo group
BOLD signal levels during fMRI n-back task | 3-6 hours after single dose of drug or placebo.
  BOLD signal level in prior regions of interest during the task (dorsolateral prefrontal cortex; hippocampus; anterior cingulate cortex) in pilosant group compared with the placebo group

SECONDARY OUTCOMES:
Optimal choice selection during loss and reward conditions in Probabilistic Instrumental Learning Task (PILT) | 3-6 hours after single dose of drug or placebo.
  Optimal choice selection during loss and reward conditions in Probabilistic Instrumental Learning Task (PILT) in pilosant group compared with the placebo group
Number of inhibited 'no-go' responses during the affective Interference Go/No-Go Task performance | 3-6 hours after single dose of drug or placebo.
  Number of inhibited 'no-go' responses during the affective Interference Go/No-Go Task in pilosant group compared with the placebo group
Accuracy of target selection on the Colour Change Detection Task | 3-6 hours after single dose of drug or placebo.
  Accuracy of target selection on the Colour Change Detection Task in pilosant group compared with the placebo group
Accuracy of emotional labeling of facial expressions during the facial emotion recognition task | 3-6 hours after single dose of drug or placebo.
  Accuracy of emotion labels (e.g. disgusted face) assigned by participants to expressive faces during the facial emotion recognition task in pilosant group compared with the placebo group
Accuracy of target selection during n-back fMRI task | 3-6 hours after single dose of drug or placebo.
  Accuracy of target selection during n-back fMRI task in pilosant group compared with the placebo group
Accuracy of stimuli labeling (novel or familiar) during fMRI memory encoding task | 3-6 hours after single dose of drug or placebo.
  Accuracy of stimuli labeling (novel or familiar) during fMRI memory encoding task in pilosant group compared with the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Susannah E Murphy, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data which has been fully de-identified may be shared with other academic and commercial organisations in the future, including those outside of the UK and the EU. Participants will be informed of this and specific consent to this is obtained within the Informed Consent Form.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: A few months after all data has been completed (ETA July 2024), unblinding has occurred (ETA April 2024), and all data analyses has been completed (ETA May 2024).
Access Criteria: The data will be made publicly available. Access requests will not be required.
URL: https://osf.io/4ckdq/

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT05849675/Prot_000.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT05849675/ICF_001.pdf